CLINICAL TRIAL: NCT03566641
Title: A Comparison of Negative Pressure Wound Therapy vs Standard Care, for Vascular, Plastic and General Surgery
Brief Title: Negative Pressure Wound Therapy vs Standard Care Dressing
Acronym: Prevena
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not start, can not secure the products.
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Munier Nazzal, M.S. M.D, Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prevena V. 11/14/17
Record Dates: First submitted 2018-04-25; First posted 2018-06-25 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Negative-Pressure Wound Therapy
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Comparing the rate of occurrence of surgical site infection, total hospital cost and length of stay between two groups: group 1 represents patients who receive Prevena for postoperative wound care and group 2 represents patients who receive standard care dressing for the same purpose.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Out study is a single-blinded randomized clinical trial. The patient will be informed about the type of dressing used for their wound care, but the investigator and the outcome assessor will be blinded for which type of dressing used for each participant patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative pressure wound therapy (Experimental): This group of patients will receive negative pressure wound therapy (prevena) as their postoperative wound care method.
  Interventions: Device: Negative pressure wound therapy
- standard care dressing (Active Comparator): This group of patients will receive standard care dressing as their postoperative wound care method.
  Interventions: Other: standard care dressing

INTERVENTIONS:
Device: Negative pressure wound therapy — The application of a vacuum across the surface of a wound through a foam dressing cut to fit the wound.
  Other Names: Prevena
  Arms: Negative pressure wound therapy
Other: standard care dressing — The application of a standard care dressing (instead of negative pressure wound therapy) across the surface of wound.
  Other Names: dray gauze
  Arms: standard care dressing

SUMMARY:
A comparison between the efficacy of negative pressure wound therapy and the efficacy of standard care dressing

DETAILED DESCRIPTION:
The aim of our study is to compare the efficacy of negative pressure wound therapy (Prevena) and standard clinical dressing in terms of prevention of postoperative surgical site infection, length of hospital stay, and total cost of hospitalization among vascular, plastic and general surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Consent for participation from the patient or his legal representative

Exclusion Criteria:

* Currently infected wounds
* Patients with history of immunosupression
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30-day postoperative period
  The rate of occurrence of signs and symptoms of surgical site infection

SECONDARY OUTCOMES:
length of total hospital stay | 6 months
  number of days of patients hospital stay after the surgery
cost of hospitalization | 6 months
  The total cost in USD of patient's hospitalization
Rate of reoperation | 30-day postoperative period
  The rate of patients' re-operation after the principal operation

CONTACTS AND LOCATIONS:
Overall Officials: munier nazzal, md, Principal Investigator — UTMC
Locations (1):
- UTMC, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No